CLINICAL TRIAL: NCT05472974
Title: Prevention of Pressure Ulcers in Patients at Medium to High Risk of Developing Pressure Ulcers and Using the DOMUS 4 / AUTO Motorized Air Mattress: Non-interventional Study
Brief Title: Prevention of Pressure Ulcers in Patients at Medium to High Risk of Developing Pressure Ulcers and Using the DOMUS 4 / AUTO Motorized Air Mattress
Status: Completed | Type: Observational
Sponsor: Wellell France (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-A01274-51
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Pressure Injury
Keywords: Pressure injury; Life support system; Beds; Prevention
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Use of a powered alternating pressure air mattress — Patients with a medium to high risk of pressure injury, without pressure injury, up during the day, will ly a on a specific P-APAM (DOMUS 4 /AUTO)

SUMMARY:
The aim of the study is to determine the clinical value of using a powered alternating pressure air mattress (P-APAM) in the prevention of pressure injury (PI) in patients at medium to high risk.

This study is noncomparative, observational study.

Patients older than 18 years of age, with a medium to high risk of PI, without PI, up during the day, and lying more than 15 hours a day on a specific P-APAM were included. The study was conducted in nursing homes, and in long-stay geriatrics department.

Patients are followed up for 35 days. The use of the P-APAM is associated with the usual PI prevention measures. The primary outcome is the percentage of patients who developed between day 0 and day 35 at least one PI of at least stage 2 on the sacrum, spine, or heel. Secondary endpoints are patient assessments of comfort, caregiver satisfaction, mattress noise level, and mattress safety.

ELIGIBILITY:
Inclusion Criteria:

Patient over 18 years old

* Patient with a medium to high risk of developing pressure ulcers (clinical judgment and a score of [10 to 14] on the Braden scale (6 (maximum risk) to 23 (no risk))
* Patient without pressure injury on the day of inclusion
* Patient up during the day, lying between 3 p.m. and 8 p.m. a day on a Domus 4 / AUTO mattress
* Patient with a weight < 200 kg
* Patient (or a trusted third party) having been informed of the study and agreeing to participate

Exclusion Criteria:

* Patient at end of life (estimated life expectancy less than 6 months)
* Malnourished patient according to the french health authority (Haute Autorité de la santé) definition*

  * For adults under 70:
  * weight loss ≥ 5% in one month or ≥ 10% in six months
  * or body mass index (BMI) ≤ 18.5 (excluding constitutional thinness)
* for adults over 70:

  * weight loss ≥ 5% in one month or ≥ 10% in six months
  * or BMI ≤ 21
  * or Mini Nutritional Assessment (MNA) ≤ 17 (/30)
  * or albuminemia < 35 g/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in nursing homes or long-stay geriatrics department
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
percentage of patients who developed at least one stage 2 pressure injury | 35 days after installation on the mattress (at day 35)
  Percentage of patients who developed at least one stage 2 PI of the sacrum, backbone, or heel (areas of support when lying down)

SECONDARY OUTCOMES:
Percentage of patients who developed a o pressure injury (any stage), other than those of the sacrum, backbone, or heel between | 35 days after installation on the mattress (at day 35)
Assessment by the patient (or family or staff in the case of incapacity) of the comfort of the mattress (general comfort, stability) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment by the nursing staff with the use of the mattress (implementation, cleaning maintenance turning, changing to a sitting position) | 35 days after installation on the mattress (at day 35)
  On a scale from 0 (not satisfied at all) to 4 (very satisfied)
Assessment of the degree of maceration | 35 days after installation on the mattress (at day 35)
  On a scale from 1 (constantly moist) to 4 rarely moist
Assessment of mattress safety | At day 35
  by collecting any adverse event or mattress malfunction during the follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie MEAUME, Pr, Principal Investigator — Hôpital ROTSCHILD
Locations (5):
- France (5):
  - Ehpad Du Parc Chateau D'Abondant, Abondant
  - Ehpad Esbv, Baugé-en-Anjou
  - Ehpad Residence Le Parc, Fontenay-aux-Roses
  - Ehpad Duc de Lorge, Saint-Jean-d'Illac
  - Ehpad Villa Du Tertre, Saint-Parres-aux-Tertres

IPD SHARING:
Plan to Share IPD: No